CLINICAL TRIAL: NCT02769598
Title: Pain Management in Pediatric Intensive Care by Studying the Autonomic Balance: Interest of Pain Hetero-assessment by Coupling ANI-HRV-scales : ANI-DOL Study
Brief Title: Pain Management in Pediatric Intensive Care by Studying the Autonomic Balance
Acronym: ANI-DOL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1500012; 1956629 (Other: CNIL)
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Pain Measurement; Children; Child, Hospitalized
Keywords: Pain; Nociception; Pediatric intensive care; Pain assessment scale; ANI index
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ANI Index for Hospitalized children: Each child will be registered upon arrival in the service and for a period of 24 hours. Registration will finish at the end of 24 hours or when the patient is discharged from the service. A FLACC scale (Face, Legs, Activity, Cry, Consolability scale) will be performed at the patient's input and then once every 4 hours corresponding to the patient's baseline. A FLACC scale will then be performed at each painful episode of the patient and 30 minutes after the end of production of analgesic treatment corresponding to the post-treatment painful condition of the patient.
  A measurement of blood pressure will be performed at each pain rating by the patient assisted by the nurse.
  Interventions: Device: ANI Index for Hospitalized children

INTERVENTIONS:
Device: ANI Index for Hospitalized children — Each file consists of a simultaneous recording of an ECG signal, according to usual practice, coupled with a record of ANI Index (Analgesia Nociception Index) by MetroDoloris®. The ECG signals and the ANI index are recorded simultaneously on a computer.
  Other Names: ANI Index

SUMMARY:
Fighting against the pain caused by the disease or by the diagnostic and therapeutic procedures for children is a daily and essential concern of health care in the pediatric sector. The quantification of pain is needed to effectively adjust analgesic therapy while limiting the side effects of treatment. Nowadays many scales are validated for children, but they are based on one-off measures and hetero assessments are often subjective and dependent on many factors including the presence of staff to children's sides.

Recent developments in the analysis of the cardiac signal in real time under the influence of autonomic control, have led to the development of a new painful stress quantification index. A monitor has recently been developed and provides an index of nociception and analgesia (ANI index). The validation of this nociception index has not been validated for pediatric care in a sector where particular attention is given to control pain.

The main purpose of this study is to show the consistency of the index compared to a validated pain scale and used routinely in non-sedated children hospitalized in pediatric intensive care units. The caregiver will have the opportunity to fine tune the effective treatment.

DETAILED DESCRIPTION:
Fighting against the pain caused by the disease or by the diagnostic and therapeutic procedures for children is a daily and essential concern of health care in the pediatric sector. The quantification of pain is needed to effectively adjust analgesic therapy while limiting the side effects of treatment. Nowadays many scales are validated for children, but they are based on one-off measures and hetero assessments are often subjective and dependent on many factors including the presence of staff to children's sides.

Recent developments in the analysis of the cardiac signal in real time under the influence of autonomic control, have led to the development of a new painful stress quantification index. A monitor has recently been developed and provides an index of nociception and analgesia (ANI index). It is based on the study of the variability of the heart rate control changes in sympathetic and parasympathetic systems in response to stimuli. Clinical correlations have been completed for most of adult patients during or after general anesthesia. The validation of this nociception index has not been validated for pediatric care in a sector where particular attention is given to control pain.

The main purpose of this study is to show the consistency of the index compared to a validated pain scale and used routinely in non-sedated children hospitalized in pediatric intensive care units. This study is based on a real-time analysis of the perception of pain in children. It is a critical validation step that could dramatically change the treatment of pediatric patients in intensive care and pediatric intensive care units by facilitating real-time patient management. The caregiver will have the opportunity to fine tune the effective treatment. The validation of this stool will allow the pain measure for children highly sedated or presenting a neuromotor handicap.

ELIGIBILITY:
Inclusion Criteria:

- Children hospitalized in pediatric intensive-care unit of the University Hospital of Saint-Etienne, painful and receiving analgesic treatment of level 2 or 3.

Exclusion Criteria:

* Children in therapy or neurological coma,
* Children enjoying a treatment known to change the ortho or parasympathetic system.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will involve 30 children aged between 2 to 18 years old who are not sedated, hospitalized in the pediatric intensive-care unit of the University Hospital of Saint-Etienne. They are expected to express an acute sensation of pain. This pain can be the result of a surgical procedure, a diagnostic or therapeutic procedure or a condition known as painful. All children studied benefit from analgesic treatment levels 2 or higher.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
ANI Index | 24 hours
  ANI Index will be measured during 24 hours and coated from 0 to 100 to have an idea of the patient's pain. It will also be compared to the FLACC Score (Face-Legs-Activity-Cry-Consolability Score) that is routinely measured and coated from 0 to 10.

SECONDARY OUTCOMES:
HFnu Index | 24 hours
  High Standard Frequency Index (HFnu) of Short Term RR variability in heart rate (HRV) in the frequency domain will be measured at 24 hours.
Ptot | 24 hours
  Ptot is a cardiac frequency variability index and it will be measured at 24 hours.
VLF | 24 hours
  VLF (Very Low Frequencies) is a cardiac frequency variability index and it will be measured at 24 hours.
LF | 24 hours
  LF (Low frequencies) is a cardiac frequency variability index and it will be measured at 24 hours.
HF | 24 hours
  HF (High Frequencies) is a cardiac frequency variability index and it will be measured at 24 hours.
LF/HF Ratio | 24 hours
  LF (Low Frequencies) / HF (High Frequencies) Ratio is a cardiac frequency variability index and it will be measured at 24 hours.
SDNN | 24 hours
  SDNN (Standard Deviation of all NN intervals) is a cardiac frequency variability index and it will be measured at 24 hours.
SDANN | 24 hours
  SDANN (Standard Deviation of the Averages of NN intervals) is a cardiac frequency variability index and it will be measured at 24 hours.
pNN50 | 24 hours
  pNN50 (NN50 count divided by the total number of all NN intervals) is a cardiac frequency variability index and it will be measured at 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No